CLINICAL TRIAL: NCT01333475
Title: Pilot Study of the Combination of MK-2206, an AKT Inhibitor, and AZD6244, a MEK Inhibitor, in Patients With Advanced Colorectal Carcinoma
Brief Title: MK-2206 and AZD6244 in Patients With Advanced Colorectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shivaani Kummar, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110117; 11-C-0117
Record Dates: First submitted 2011-04-09; First posted 2011-04-12 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2014-11

CONDITIONS: Colorectal Neoplasms
Keywords: Targeted Therapy; KRAS Mutation; Metastatic Colorectal Cancer; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — MK 2206; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAC1:MK-2206 & AZD6244 in Pts with Colorectal Ca (Experimental): Cycle = 28 days:MK-2206:90 mg PO days 1, 8, 15, and 22 AZD6244 Hydrogen sulfate: 75 mg PO QD (every day) MK-2206 + AZD6244: MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression.
  Interventions: Drug: MK-2206 + AZD6244
- TAC1A:MK-2206 & AZD6244 in Pts with Colorectal Ca (Experimental): Cycle = 28 days:MK-2206:135 mg PO days 1, 8, 15, and 22 AZD6244 Hydrogen sulfate: 100 mg PO QD
  MK-2206 + AZD6244: MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression.
  Interventions: Drug: MK-2206 + AZD6244

INTERVENTIONS:
Drug: MK-2206 + AZD6244 — MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression.

SUMMARY:
Background:

- MK-2206 and AZD6244 (Selumetinib) are experimental cancer treatment drugs that block the effect of certain proteins that cancer cells need to grow and survive. These drugs may be effective treatments for some types of colorectal cancer that has not responded to or has relapsed after standard treatment. Researchers are interested in studying how MK-2206 and AZD6244 affect levels of certain proteins in colorectal cancer tumor, and how well the drugs work against cancer cells by examining cells from a tumor sample collected before the drugs are given and again after the drugs are given.

Objectives:

- To evaluate the safety and effectiveness of MK-2206 and AZD6244 in individuals with advanced colorectal carcinoma that has not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with advanced colorectal carcinoma that has not responded to at least one type of standard chemotherapy.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and tumor imaging studies.
* Participants will take MK-2206 and AZD6244 by mouth for 4-week cycles of treatment, with one dose of MK-2206 per week and one dose of AZD6244 every day. (If participants have negative side effects from the medications, the doses will be adjusted to a smaller dose). Participants will keep a diary to record doses and keep track of any side effects.
* During treatment, participants will have regular visits to the clinical center, involving blood and urine tests, tumor biopsies, and other examinations to monitor the effects of treatment. Participants will have imaging studies every two cycles (8 weeks) to study the cancer's response to the treatment.
* Participants will continue to have cycles of treatment for as long as the treatment continues to be effective and the side effects are not severe enough to stop participation in the study....

DETAILED DESCRIPTION:
Background:

* The PI3K-AKT (protein kinase B) and RAF/MEK (methyl ethyl ketone)/ERK (extracellular-signal regulated kinase) pathways are two of the most frequently activated signaling pathways in cancer, including colorectal cancer (CRC). KRAS (Kirsten Rat Sarcoma Viral Oncogene Homolog) mutations are detected in approximately 40% of patients with CRC and predict for resistance to EGFR (epidermal growth factor receptor) inhibitors. AKT is upregulated in approximately 60% of CRC.
* Preclinical studies demonstrate that activating mutations in the PI3K-AKT pathway and increased phosphorylated Akt through a MEK-EGFR-PI3K feedback loop are implicated in resistance to the antitumor effect of MEK inhibition.
* MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS (Rat Sarcoma) pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression. The combination is being studied in a Phase I trial and appears tolerable.

Primary Objectives:

* Determine reduction of pERK and pAKT in tumor biopsies on C1D1 (cycle 1 day 1) post-administration of the combination of AZD6244 hydrogen sulfate and MK-2206 in patients with advanced colorectal cancer, stratified for KRAS mutation status.
* Evaluate for recovery of pAKT levels in tumor biopsy samples obtained on C1D4 (cycle 1, day 4) after administration of the combination of AZD6244 hydrogen sulfate and MK-2206 in patients with advanced colorectal cancer, stratified for KRAS mutation status.
* Determine reduction of Ki-67 in tumor biopsies post-administration of the combination of AZD6244 hydrogen sulfate and MK-2206 in patients with advanced colorectal cancer, stratified for KRAS mutation status.

Secondary Objectives:

* Evaluate reduction of pERK and pAKT in peripheral blood mononuclear cells (PBMCs) after administration of the combination of AZD6244 hydrogen sulfate and MK-2206 and correlate these reductions with those seen in tumor biopsy samples.
* Evaluate antitumor activity of the combination of MK-2206 with AZD6244 hydrogen sulfate.

Eligibility:

-Patients with histologically documented colorectal cancer that has progressed or recurred after oxaliplatin- and irinotecan-based chemotherapy for metastatic disease. KRAS mutation analysis results must be available prior to enrollment. Patients must have disease amenable to biopsy, and be willing to undergo pre-and post-treatment tumor biopsies.

Study Design:

* MK-2206 135 mg PO (by mouth) once weekly and AZD6244 hydrogen sulfate 100 mg PO (by mouth) once daily will be administered in 28-day cycles, beginning on C1D1 (cycle 1, day 1).
* Patients will be stratified for KRAS mutation status.
* Blood samples and paired mandatory tumor biopsies will be obtained for pharmacodynamic studies.
* CT (computed tomography) scans will be performed every 2 cycles for restaging.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed metastatic colorectal cancer, which has recurred or progressed following oxaliplatin- and irinotecan-based chemotherapy regimens administered for the treatment of metastatic disease, except if the patient was not a candidate for either agent or refused treatment with oxaliplatin or irinotecan. The diagnosis must be confirmed by the Laboratory of Pathology at the Clinical Center, NIH (National Institutes of Health), prior to patient enrollment.
* Results of KRAS (Kirsten-Ras) mutation analysis must be available prior to patient enrollment.
* Patients must have disease amenable to biopsy, and must be willing to undergo pre- and post-treatment tumor biopsies.
* Patients must have completed any major surgery chemotherapy, radiation therapy, or biologic therapy greater than or equal to 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin C). Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in an exploratory IND (investigational new drug) /Phase 0 study. Patients must have recovered to eligibility levels from any prior surgery, toxicity, or adverse events.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of MK-2206 in combination with AZD6244 in patients less than 18 years of age, children are excluded from this study.
* Life expectancy of greater than 3 months.
* ECOG (Eastern Cooperative Oncology Group) performance status less than 2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/microL
  * Platelets greater than or equal to 100,000/microL
  * Total bilirubin less than or equal to 1.5 times institutional ULN (upper limit of normal)
  * AST (aspartate aminotransferase) /ALT (alanine aminotransferase) less than or equal to 3.0 times institutional ULN; less than or equal to 5.0 times institutional ULN if liver metastases
  * Creatinine less than 1.5 times ULN; OR
  * Measured creatinine greater than or equal to 60 mL/minute for patients with clearance creatinine levels greater than or equal to 1.5 times ULN
  * INR (International Normalized Ratio) less than or equal to 1.4
  * PTT (partial thromboplastin time) less than or equal to 40 seconds unless due to lupus anticoagulant
* The effects of MK-2206 and of AZD6244 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 weeks after dosing with study medication ceases. However, adequate contraception for male patients should be used for 16 weeks post- last dose due to sperm life cycle. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of child-bearing potential must have a negative pregnancy test prior to entry.
* Patients must be able to swallow whole tablets and capsules. Tablets must not be crushed or chewed; capsules must not be opened.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 4 weeks after treatment of the brain metastases, without steroids. Patients on stable doses of antiseizure medications with no history of seizures in the past 4 weeks will be eligible.
* Poorly controlled diabetes defined as fasting blood glucose of greater than 160 mg/dL (CTCAE (Common Terminology Criteria for Adverse Events)) Grade greater than or equal to 2) or HgA1c (glycated hemoglobin) greater than 8%.
* QTc (corrected QT interval) prolongation greater than 450 msec (male) or QTc greater than 470 msec (female) by Bazetts formula or use of medications that may cause QTc interval prolongation. A comprehensive list of agents with the potential to cause QTc prolongation can be found at http://www.azcert.org/medical-pros/drug- lists/bycategory.cfm.
* Patients with clinically significant intercurrent illnesses, including but not limited to, interstitial pneumonitis, pulmonary fibrosis, uncontrolled infection, psychiatric illness or social situations that would limit compliance with study requirements.
* Patients with symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, myocardial infarction in the past 6 months, left ventricular ejection fraction (LVEF) less than or equal to 50%, are not eligible to participate.
* Uncontrolled hypertension (blood pressure [BP] of greater than or equal to 150/95 despite optimal therapy).
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
* HIV (human immunodeficiency virus) -positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MK-2206 and AZD6244.
* Patients currently on warfarin (Coumadin) are ineligible. Otherwise eligible patients requiring anticoagulant treatment should have their warfarin switched to a low molecular weight heparin such as enoxaparin injections.
* Patients on strong cytochrome P450 system inducers or inhibitors are ineligible.

INCLUSION OF WOMEN AND MINORITIES:

-Both men and women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Messa C, Russo F, Caruso MG, Di Leo A. EGF, TGF-alpha, and EGF-R in human colorectal adenocarcinoma. Acta Oncol. 1998;37(3):285-9. doi: 10.1080/028418698429595. PMID 9677101
- [Background] Cunningham D, Humblet Y, Siena S, Khayat D, Bleiberg H, Santoro A, Bets D, Mueser M, Harstrick A, Verslype C, Chau I, Van Cutsem E. Cetuximab monotherapy and cetuximab plus irinotecan in irinotecan-refractory metastatic colorectal cancer. N Engl J Med. 2004 Jul 22;351(4):337-45. doi: 10.1056/NEJMoa033025. PMID 15269313
- [Background] Khosravi-Far R, Der CJ. The Ras signal transduction pathway. Cancer Metastasis Rev. 1994 Mar;13(1):67-89. doi: 10.1007/BF00690419. PMID 8143346
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0117.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because dual target evaluation of >70% was not observed in the tumor biopsies from any of the participants evaluated, no participants were enrolled to Cohort C to evaluate target recovery.
  TAC1 and TAC1A -Since all patients received both drugs, each of the TACs (Treatment Assignment Code) reflect the dose level.
Groups:
- TAC1: Cycle = 28 days:MK-2206:90 mg PO days 1, 8, 15, and 22 AZD6244 Hydrogen sulfate: 75 mg PO QD
  MK-2206 + AZD6244: MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression.
- TAC1A: Cycle = 28 days:MK-2206:135 mg PO days 1, 8, 15, and 22 AZD6244 Hydrogen sulfate: 100 mg PO QD
  MK-2206 + AZD6244: MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression.
Period: Overall Study
Arm/Group | TAC1 | TAC1A
Started | 12 | 9
Completed | 10 | 6
Not Completed | 2 | 3
Not completed — pt withdrew-need emergent radiation trmt | 1 | 0
Not completed — Toxicity | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- TAC1A: Cycle = 28 days:MK-2206: 135 mg PO days 1, 8, 15, and 22 AZD6244 Hydrogen sulfate: 100 mg PO QD
  MK-2206 + AZD6244: MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression.
- Total: Total of all reporting groups
Arm/Group | TAC1 | TAC1A | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (16.4) | 53.8 (9.3) | 54.0 (13.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — One participant selected White and Asian for Race, thus the category "More than one race" was selected. Six participants versus seven is noted in the "White" category and no participants is noted in the "Asian" category.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 10 | 6 | 16
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 8 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: pERK and pAKT Levels in Tumor Biopsies on C1D1 and C1D22 Post-administration of the Combination of AZD6244 Hydrogen Sulfate and MK-2206 in Participants With Advanced Colorectal Cancer
Description: A predetermined target inhibition reduction of 70% of both pERK and pAKT was deemed significant, thus tumor biopsies were performed at C1D1 or C1D22 post administration and evaluated using quantitative chemiluminescence immunoassay to measure pERK and pAKT levels in human tissue.
Time Frame: C1D1 and C1D22 post administration of the combination of AZD6244 hydrogen sulfate and MK-2206
Measure: Mean (Full Range); unit: pg/ µg of protein
Groups:
- TAC1A: Cycle = 28 days:MK-2206: 135mg PO days 1, 8, 15, and 22 AZD6244 Hydrogen sulfate: 100 mg PO QD
  MK-2206 + AZD6244: MK-2206 and AZD6244 hydrogen sulfate are selective inhibitors of human AKT and MEK, respectively, with preclinical and clinical anti-tumor activity as single agents and in combination with a variety of drugs. Combination treatment in mouse cancer models harboring mutations in both the PI3K and RAS pathways was more potent compared to either agent used alone, and resulted in substantial tumor inhibition, including tumor regression.
Arm/Group | TAC1 | TAC1A
Number analyzed (Participants) | 10 | 6
pg/ µg of protein
  pAKT Baseline C1D1 | 4.86 [1.89 to 7.41] | 0 [0 to 0]
  pAKT post administration C1D1 | 2.20 [1.44 to 3.44] | NA [NA to NA] — N/A values identify levels that were not investigated - no participants were enrolled.
  pAKT Baseline C1D22 | NA [NA to NA] — N/A values identify levels that were not investigated - no participants were enrolled. | 4.22 [1.56 to 7.64]
  pAKT Post administration C1D22 | NA [NA to NA] — N/A values identify levels that were not investigated - no participants were enrolled. | 2.91 [1.27 to 7.3]
  pERK Baseline C1D1 | 5.06 [1.56 to 12.26] | NA [NA to NA] — N/A values identify levels that were not investigated - no participants were enrolled.
  pERK post administration C1D1 | 2.77 [1.56 to 4.93] | NA [NA to NA] — N/A values identify levels that were not investigated - no participants were enrolled.
  pERK Baseline C1D22 | NA [NA to NA] — N/A values identify levels that were not investigated - no participants were enrolled. | 3.97 [1.56 to 7.19]
  pERK Post administration C1D22 | NA [NA to NA] — N/A values identify levels that were not investigated - no participants were enrolled. | 3.5 [1.56 to 6.82]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: 29 months, 23 days
Measure: Number; unit: participants
Arm/Group | TAC1 | TAC1A
Number analyzed (Participants) | 12 | 9
participants | 12 | 8

ADVERSE EVENTS:
Arm/Group | TAC1 | TAC1A
Serious Adverse Events (participants affected / at risk) | 5/12 | 6/9
Other Adverse Events (participants affected / at risk) | 12/12 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAC1 (N=12) | TAC1A (N=9)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) — progressive disease
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) — progressive disease; disease progression
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) — tumor resection
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAC1 (N=12) | TAC1A (N=9)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 3 (4)
Alanine aminotransferase increased (Investigations) | 7 (16) | 6 (11)
Alkaline phosphatase increased (Investigations) | 7 (16) | 6 (9)
Allergic rhinitis (Immune system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (11) | 4 (11)
Anorexia (Metabolism and nutrition disorders) | 3 (5) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (27) | 5 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Bloating (Gastrointestinal disorders) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 5 (9) | 1 (1)
Blurred vision (Eye disorders) | 1 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CPK increased (Investigations) | 4 (6) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (5) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (9) | 4 (11)
Dizziness (Nervous system disorders) | 2 (2) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 1 (3)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (9) | 2 (2)
Fever (General disorders) | 1 (1) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (10) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (15) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 10 (39) | 7 (22)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (24) | 6 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (11) | 2 (5)
Hyponatremia (Metabolism and nutrition disorders) | 7 (9) | 4 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) — infection limbs
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — small intestine
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — right small toe bruising/laceration
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (11) | 6 (11)
Lymphocyte count increased (Investigations) | 1 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (13) | 5 (14)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 3 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) — night dreams
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (2) — vivid dreams
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — dry nose
Retinal detachment (Eye disorders) | 4 (4) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (10) | 4 (11)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No